CLINICAL TRIAL: NCT01436331
Title: A Pragmatic Cluster Randomized Controlled Trial of a Multi-element Psychosocial Intervention for Early Psychosis in a 10 Million Inhabitant Catchment Area Aimed to Measure the Treatment's Feasibility and Effectiveness: GET UP-PIANO Trial
Brief Title: A Large Pragmatic Cluster Randomized Controlled Trial of a Multi-element Psychosocial Intervention for Early Psychosis
Acronym: GETUP-PIANO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Ruggeri, Mirella, Professor of Psychiatry, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1682; C.U.P. H 61J08000200001 (Other: Veneto Region - Italy)
Record Dates: First submitted 2011-09-14; First posted 2011-09-19 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Psychosis
Keywords: First episode psychosis; Early Psychosis; Cognitive Behavioural therapy; Psychosocial Intervention; Assertive Community treatment; Family Intervention; Mental Disorders; Psychotic Disorders; Schizophrenia and Disorders with Psychotic Features; Affective Disorders, Psychotic
MeSH Terms: conditions — Psychotic Disorders; Mental Disorders; Schizophrenia Spectrum and Other Psychotic Disorders; Affective Disorders, Psychotic | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment As Usual (TAU) (Active Comparator)
  Interventions: Other: Treatment As Usual (TAU)
- TAU+CBT for pts+Family Intervention+CM (Experimental)
  Interventions: Behavioral: TAU+CBT for pts+Family Intervention+CM.

INTERVENTIONS:
Other: Treatment As Usual (TAU) — Services participating in the trial are routine public Community Mental Health Centres (CMHCs), which operate within the Italian National Health Service. Multi-disciplinary teams operating these CMHCs provide a wide range of integrated programmes, including inpatient care, day care, rehabilitation, outpatient care, home visits, 24-hour emergency services, and residential facilities. Standard care for FEP patients generally consists of personalized outpatient psychopharmacological treatment, combined with non-specific supportive clinical management at the CMHC level. Family interventions generally consist of non-specific informal support/educational sessions. Both specialized individual psychotherapeutic interventions for patients (included CBT) and specialized psycho-educational or cognitive-oriented family interventions are usually not provided, due to lack of trained professionals.
  Other Names: standard treatment; control treatment
  Arms: Treatment As Usual (TAU)
Behavioral: TAU+CBT for pts+Family Intervention+CM. — The experimental treatment package is administered by the CMHC staff, after training and with ongoing supervision by experts. Cognitive-behavioural therapy (CBT) is based on the model developed by Kuipers in 1998 and Garety in 2008. A total of 20-30 CBT sessions per patient will be delivered, with weekly sessions during months 1-3 and fortnightly over the following 6 months. Family Intervention is based on the model proposed by Leff in 1982 and further developed by Kuipers in 2002. It includes a total of 10-15 sessions with each individual family: 6 in months 1-3, and at least 1 session/month in the 6 months afterwards. Every patient/family will have a dedicated Case Manager, who will coordinate all planned interventions. Specific training programs have been developed, with assessment of the staff competence. Detailed Manuals based on international standards have been developed and will be used. Fidelity will be measured at the end of the trial.
  Other Names: Multi-element intervention; Family psychoeducation
  Arms: TAU+CBT for pts+Family Intervention+CM

SUMMARY:
Multi-element interventions for first-episode psychosis (FEP) are promising but have mostly been conducted on non epidemiologically representative samples in experimental settings, raising the risk thereby of underestimating the complexities involved in treating onset psychosis in "real world" services. The PIANO Trial (Psychosis early Intervention and Assessment of Needs and Outcome) is part of a more broad-based research program (Genetics, Endophenotype and Treatment: Understanding early Psychosis - GET UP) and aims to: 1) test, at 9 months, the effectiveness, as compared to treatment as usual (TAU) of multi-component psychosocial intervention on a large epidemiologically-based cohort of FEP patients and their family members recruited from a 10 million inhabitant catchment area; 2) identify barriers that may hinder its feasibility and patient/family conditions that can render this type of treatment ineffective or inappropriate; 3) identify clinical, psychological, and environmental and service predictors of treatment effectiveness in FEP.

Study participants will be recruited from Community Mental Health Centers (CMHCs) operating for the Italian National Health Service and located in several Northern and Central Regions of Italy. The GET UP PIANO Trial has a pragmatic cluster randomized controlled design, which is considered the gold standard approach for trials that evaluate complex interventions implemented at the institutional level, with the aim of improving health. The assignment units (clusters) are the CMHCs, and the units of observation and analysis are the Centers' patients and their family members.

Patients in the experimental group will receive TAU plus: (a) Cognitive-Behavioural Therapy (CBT) sessions, (b) psycho-educational sessions for family members, and c) a case manager, to serve as the patient's referent. Patient enrollment will take place over a 1 year interval, after a 3 month-long piloting. The fidelity of the experimental interventions and the characteristics of TAU will be regularly monitored. Several psychopathological, psychological, functioning and service use variables will be assessed at baseline and 9 month follow-up by independent evaluators. Assuming an expected incidence rate of 17/100.000 per year for functional psychoses (as previously estimated in Italy), the investigators expect to recruit about 800 patients, and 600 relatives. Assuming an attrition rate of about 50%, the size of the trial would detect at 9 months a difference in terms of primary outcome from 25% for the TAU arm to 10% for the intervention arm, with a power of 80%.

DETAILED DESCRIPTION:
BACKGROUND. It has been shown that most clinical and psychosocial deterioration in psychosis occurs within the first 5 years of illness onset, suggesting thereby that this timeframe is a "critical" period for initiating treatment. Research has therefore more recently focused on early detection and intervention for psychosis, showing that the beneficial effects of antipsychotic medication on first-episode psychosis (FEP) are tempered by the fact that, despite initial symptom reduction, functional recovery is typically poor, even when optimal pharmacological treatment is provided. Family members suffer due to the high emotional burden of being caregivers and frequently show signs of psychological distress. Over the last few years, there has been a growing interest in psychosocial intervention as a means of facilitating recovery and reducing long-term disability associated with psychosis. Literature on psychosocial interventions in FEP can be viewed in terms of two broad categories: 1) studies evaluating specific (i.e. single-element) psychosocial interventions (e.g. individual cognitive behavioral therapy), and 2) studies evaluating comprehensive (i.e. multi-element) interventions, which may include early detection strategies, individual, group, and/or family therapy, and case management (in addition to pharmacological treatment). The latter appear very promising and have been found to be associated with symptom reduction/remission, improved quality of life, increased social and cognitive functioning, low inpatient admission rates, improved insight, high degree of satisfaction with treatment, less time spent in hospital, decreased substance abuse, and fewer self- harm episodes. Most multi-element research programs, however, have been conducted on non-epidemiologically representative samples in experimental settings, raising the risk thereby of underestimating the complexities involved in treating FEP in "real world" services. Moreover, these interventions have rarely tested their efficacy against a control group or, if they have done so, they have used historical or prospective comparison groups, or single-group designs, which track the progress of a single group over a given period of time. With respect to practices, over the last 10 years, some countries have implemented specific early psychosis interventions, but even these have not yet become routinely conducted. Few studies have identified barriers that can hinder the feasibility of these interventions or the pinpointing of patient or family conditions that can render this type of ineffective or inappropriate. Hence, efforts to implement these specific multi-element interventions should be accompanied by rigorous scientific methodology, with the aim of better understanding the actual effectiveness of this approach.

AIMS. The PIANO Trial (Psychosis early Intervention and Assessment of Needs and Outcome described herein makes up part of the more broad-based research program Genetics Endophenotypes and Treatment: Understanding early Psychosis (GET UP, National Coordinator: Prof. Mirella Ruggeri, Verona), which is financed by the Italian Ministry of Health as part of a Ricerca Sanitaria Finalizzata and is coordinated by the Azienda Ospedaliera Universitaria Integrata in Verona. GET UP Research Programme consists of 4 partner Projects: PIANO (Psychosis: early Intervention and Assessment of Needs and Outcome); TRUMPET (TRaining and Understanding of service Models for Psychosis Early Treatment); GUITAR (Genetic data Utilization and Implementation of Targeted drug Administration in the clinical Routine); and CONTRABASS (COgnitive Neuroendophenotypes for Treatment and RehAbilitation of psychoses: Brain imaging, inflAmmation and StresS). Each of these partner projects pertains to different areas of research, but are linked together in a high degree of harmonization of effort.

The Trial described herein - which is the main component of GET UP PIANO, and the main data collection axis for the overall GET UP Research Program - aims to: 1) test, at 9 months, the effectiveness, as compared to treatment as usual (TAU) of multi-component psychosocial intervention on a large epidemiologically-based cohort of FEP patients recruited from a 10 million inhabitant catchment area; 2) verify the clinical routine limits of this approach, i.e. to identify barriers that may hinder its feasibility and patient/family conditions that can render this type of treatment ineffective or inappropriate; 3) identify clinical, psychological, and environmental and service predictors of treatment effectiveness in FEP, as undertaken in an Italian community mental health care framework.

Study participants will be recruited from Community Mental Health Centres (CMHCs) operating for the Italian National Health Service and located in several Northern and Central Regions of Italy. Specifically, the Participating Units (PU) will be located in the Veneto Region (subdivided in the Western Veneto and in the Eastern Veneto PU), the Emilia-Romagna Region (subdivided in the Emilia and Romagna PUs) and in the provinces of Florence, Bolzano, and Milano (subdivided in the Milan Niguarda and in the Milan San Paolo PUs), and thus, overall, a 10 million-inhabitant catchment area.

DESIGN. The GET UP PIANO Trial has a pragmatic cluster randomized controlled design, which compares the effectiveness of a multi-element psychosocial treatment for FEP patients and their family members, versus the treatment as usual provided by Italian community mental health services. A cluster design was chosen based on feasibility considerations. In fact, a document drafted by members of the MRC Health Services and Public Health Research Board in 2000 indicated cluster randomisation as the gold standard approach for trials that evaluate complex interventions implemented at the institutional level, with the aim of improving health. The assignment units (clusters) will be the catchment area's CMHC, and the units of observation and analysis will be the Centers' patients and their family members.

CMHCs enrollment procedure: The PIANO Trial catchment area has 126 CMHCs (9.951.306 inhabitants), all of which have been officially asked to participate in GET UP; 117 have accepted to participate, covering a catchment area of 9.304.093 inhabitants thereby. In an effort to improve the study design's efficiency, before randomization the investigators divided CMHCs into strata, according to three variables: affiliation to the same community psychiatric service, CMHC catchment area size, urban/mixed vs. rural. The socio-economic levels in the trial catchment area were found to be quite homogeneous, and the variable of urban/mixed vs. rural stratification accounted for most of the differences observed. With the exception of staff members in 5 CMHCS (covering a catchment area of 503.000 inhabitants) the mental health staff of the remaining 112 CMHCs had received no prior training in the intervention used in the trial. These first 5 Centers were therefore forced to the intervention arm, and this subgroup will be used as the expected "gold standard" in the analysis to measure the competence of the remaining professionals. Thus, 112 CMHCs (8.801.093 inhabitants) were available for the randomization procedure and were entered in the randomization procedure, with equal numbers being allocated to each arm. Based on administrative data in these Centers, the at-risk population (18-54 years) was estimated to be approximately 50% of the total inhabitants. Assuming an expected incidence rate of 17/100.000 per year for non affective and affective psychoses (as previously estimated in Italy) the investigators can expect to recruit over one year in the catchment area about 800 patients at their first episode of psychosis, and 600 relatives. Assuming an attrition rate of about 50%, the size of the trial would detect at 9 months a difference in terms of primary outcome from 25% for the TAU arm to 10% for the intervention arm, with a power of 80%.

Patient- and family member enrollment procedure: Patient enrollment will take place over a 1 year interval, after a 3 month-long piloting. Interventions begin within one month from intake, and, in any event, as soon as each patient is stabilized. Clinical stabilization is defined as a condition allowing the patient to collaborate in at least a brief examination. Patients in the experimental group will receive treatment as usual plus: (a) Cognitive Behavioural Therapy (CBT) sessions, (b) psycho-educational sessions for family members, and c) a Case Manager (CM), to serve as the patient's referent. Treatment as usual conducted in the control arm CMHSs has been characterized in previous studies. The fidelity of the experimental interventions and the characteristics of treatment as usual will be regularly monitored.

BASELINE ASSESSMENT. Before entering the study, patients screening positive for psychosis will be asked to provide informed consent to participate. When patients are considered clinically stabilized (after intake), they will be assessed by independent evaluators with a set of standardized instruments which measure: substance abuse (Clinical Drug Use Scale, CDUS), symptoms (Positive and Negative Syndrome Scale, PANSS; Hamilton Rating Scale for Depression, HAMD; Bech-Rafaelsen Mania rating Scale, BRMRS); global functioning (Global Assessment of Functioning, GAF); Subjective appraisal of positive symptoms (Psychotic Symptom Rating Scales, PSYRATS), social disability (Disability Assessment Scale, WHO-DAS), insight (Schedule for Assessment of Insight, SAI-E), needs for care (Camberwell Assessment of Need, CAN-EU), quality of life (WHO-QOL), life events (first 14 years of life, one year prior to the onset of psychosis, period following onset measured with ad hoc schedule for Life Events, CECA-Q), parental bonding (Parental Bonding Instrument,PBI), and expressed emotions (Level of Expressed Emotion Scale, LEE). Participating patients will be asked for consent to involve their family members in the trial, and when given, family members also providing informed consent will be assessed regarding burden of care (Involvement Evaluation Questionnaire, IEQ) and emotional distress (General Health Questionnaire, GHQ); they will also be interviewed with respect to the patient's pre-morbid adjustment (Pre-morbid Adjustment Scale, PAS) and obstetric complications at birth.

FOLLOW-UP ASSESSMENT. After 9 months from baseline, patients will be re-assessed for substance abuse, psychotic symptoms (PANSS and PSYRATS) depression (HAMD, BRMS), global functioning (GAF), social disability (WHO DAS), insight (SAI-E), needs for care (CAN), and quality of life (WHO-QoL). Moreover, patients will be evaluated in terms of pharmacological side effects, pattern of clinical course (Life Chart Schedule), and service satisfaction (Verona Service Satisfaction Scale-Patient version,VSSSP ). Family members will be re-assessed with respect to burden of care (IEQ) and emotional distress (GHQ); they will also be assessed for service satisfaction (VSSS-Relative version).

ELIGIBILITY:
Inclusion Criteria:

1. age 18-54 yrs
2. residence in the catchment area of participating Community Mental Health Centres
3. presence of (a) at least 1 of the following symptoms: hallucinations, delusions, qualitative speech disorder, qualitative psychomotor disorder, bizarre or grossly inappropriate behavior, or (b) at least 2 of the following symptoms: loss of interest, initiative and drive, social withdrawal, episodic severe excitement, purposeless destructiveness, overwhelming fear, marked self-neglect
4. first lifetime contact with participating CMHC, occasioned by symptoms enumerated in 3.
5. clinical ICD-10 diagnosis of F20-29; F30.2, F31.2, F31.5, F31.6, F32.3, F33.3, F1x.4; F1x.5; F1x.7;F20-F29, as confirmed after 6 months by using the Schedule for Clinical Assessment in Neuropsychiatry (WHO SCAN)

Exclusion Criteria:

1. prior anti-psychotic medication (> 3 months) provided by any psychiatric or other medical agencies
2. mental disorders due to a general medical condition

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 626 (Actual)
Dates: Start 2010-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Relapses | 9 months
  We define relapse as an episode that has resulted in an admission to a psychiatric inpatient unit (number and days of hospitalization) and/or any case noted record of increase in psychotic symptoms' severity during the study period
Positive and negative symptoms | change from baseline at 9 month follow-up
  Positive and Negative symptoms will be measured by the positive and negative subscales of the PANSS and by the PSYRATS

SECONDARY OUTCOMES:
Service Satisfaction in patients and relatives | 9 months
  Service satisfaction will be measured by using the Verona Service Satisfaction Scale, versions for patients and relatives
Patient Functioning | change from baseline at 9 month follow-up
  Functionig will be assessed by using the Global Assessment of Functioning Scale and the WHO-Disability Assessment Scale
Patient emotional wellbeing | change from baseline at 9 month follow-up
  Emotional wellbeing will be measured by using the anxiety and depression items of the PANSS and the Hamilton-D and selected items of the WHO QoL Scale
Service disengagement | 9 months
  Service disengagement and time to service disengagement will be assessed by consulting case records and local databases
Patient Needs for care | change from baseline at 9 month follow-up
  Needs for care will be assessed by using the Camberwell Assessment of Need scale
Key relative expressed emotions | change from baseline at 9 month follow-up
  Expressed emotions will be measured by using the Level of Expressed Emotion Scale
Key relative burden | change from baseline at 9 month follow-up
  Family burden will be measured by using the Involvement Evaluation Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Mirella RUGGERI, M.D., Principal Investigator — Universita' di Verona
Locations (1):
- University of Verona - Section of Psychiatry and Clinical Psychology, Department of Public Health and Community Medicine, Verona, Italy

REFERENCES:
- [Background] Brown H, Prescott R. Applied Mixed Models in Medicine. John Wiley & Sons, 1999
- [Background] Campbell MK, Mollison J, Grimshaw JM. Cluster trials in implementation research: estimation of intracluster correlation coefficients and sample size. Stat Med. 2001 Feb 15;20(3):391-9. doi: 10.1002/1097-0258(20010215)20:33.0.co;2-z. PMID 11180309
- [Background] Donner A, Klar N. Statistical considerations in the design and analysis of community intervention trials. J Clin Epidemiol. 1996 Apr;49(4):435-9. doi: 10.1016/0895-4356(95)00511-0. PMID 8621994
- [Background] Edwards J, Harris MG, Bapat S. Developing services for first-episode psychosis and the critical period. Br J Psychiatry Suppl. 2005 Aug;48:s91-7. doi: 10.1192/bjp.187.48.s91. PMID 16055816
- [Background] Eldridge S, Cryer C, Feder G, Underwood M. Sample size calculations for intervention trials in primary care randomizing by primary care group: an empirical illustration from one proposed intervention trial. Stat Med. 2001 Feb 15;20(3):367-76. doi: 10.1002/1097-0258(20010215)20:33.0.co;2-r. PMID 11180307
- [Background] Garety PA, Fowler DG, Freeman D, Bebbington P, Dunn G, Kuipers E. Cognitive--behavioural therapy and family intervention for relapse prevention and symptom reduction in psychosis: randomised controlled trial. Br J Psychiatry. 2008 Jun;192(6):412-23. doi: 10.1192/bjp.bp.107.043570. PMID 18515890
- [Background] Guittet L, Ravaud P, Giraudeau B. Planning a cluster randomized trial with unequal cluster sizes: practical issues involving continuous outcomes. BMC Med Res Methodol. 2006 Apr 12;6:17. doi: 10.1186/1471-2288-6-17. PMID 16611355
- [Background] Hahn S, Puffer S, Torgerson DJ, Watson J. Methodological bias in cluster randomised trials. BMC Med Res Methodol. 2005 Mar 2;5:10. doi: 10.1186/1471-2288-5-10. PMID 15743523
- [Background] Kerry SM, Bland JM. Unequal cluster sizes for trials in English and Welsh general practice: implications for sample size calculations. Stat Med. 2001 Feb 15;20(3):377-90. doi: 10.1002/1097-0258(20010215)20:33.0.co;2-n. PMID 11180308
- [Background] Kuipers E, Fowler D, Garety P, Chisholm D, Freeman D, Dunn G, Bebbington P, Hadley C. London-east Anglia randomised controlled trial of cognitive-behavioural therapy for psychosis. III: Follow-up and economic evaluation at 18 months. Br J Psychiatry. 1998 Jul;173:61-8. doi: 10.1192/bjp.173.1.61. PMID 9850205
- [Background] Kuipers E, Leff J, Lam D. Family work for schizophrenia: a practical guide, 2nd Edition. Gaskell:London,2002
- [Background] Leff J, Kuipers L, Berkowitz R, Eberlein-Vries R, Sturgeon D. A controlled trial of social intervention in the families of schizophrenic patients. Br J Psychiatry. 1982 Aug;141:121-34. doi: 10.1192/bjp.141.2.121. PMID 7116051
- [Background] Lora A, Corlito G, Miceli M, Di Munzio W, Lasalvia A, Tanini A, Mari L, Casacchia M, Magnani N, Cristofalo D, Semisa D, Ruggeri M; Gruppo SIEP-DIRECT'S. [The treatment of acute psychotic episode: discrepancy between routine practice and evidence. The Project SIEP-DIRECT'S]. Epidemiol Psichiatr Soc. 2008 Oct-Dec;17(4):319-30. Italian. PMID 19024720
- [Background] Murray DM. Design and Analysis of Group-Randomized Trials. Oxford University Press, 1998.
- [Background] Murray DM, Varnell SP, Blitstein JL. Design and analysis of group-randomized trials: a review of recent methodological developments. Am J Public Health. 2004 Mar;94(3):423-32. doi: 10.2105/ajph.94.3.423. PMID 14998806
- [Background] Penn DL, Waldheter EJ, Perkins DO, Mueser KT, Lieberman JA. Psychosocial treatment for first-episode psychosis: a research update. Am J Psychiatry. 2005 Dec;162(12):2220-32. doi: 10.1176/appi.ajp.162.12.2220. PMID 16330584
- [Background] Ruggeri M, Lora A, Semisa D; SIEP-DIRECT'S Group. The SIEP-DIRECT'S Project on the discrepancy between routine practice and evidence. An outline of main findings and practical implications for the future of community based mental health services. Epidemiol Psichiatr Soc. 2008 Oct-Dec;17(4):358-68. PMID 19024723
- [Background] Ruggeri M, Tansella M. Achieving a better knowledge on the causes and early course of psychoses: a profitable investment for the future? Epidemiol Psichiatr Soc. 2007 Apr-Jun;16(2):97-101. doi: 10.1017/s1121189x00004693. No abstract available. English, Italian. PMID 17619538
- [Background] Ruggeri M, Tansella M. Improving the treatment of schizophrenia in real world mental health services. Epidemiol Psichiatr Soc. 2008 Oct-Dec;17(4):249-53. No abstract available. English, Italian. PMID 19024711
- [Background] Ruggeri M, Bacigalupi M, Casacchia M, Miceli M, Morganti C, Scavo V, Allevi L, Lupoi S, Cristofalo D, Lasalvia A, Lora A, Semina D; Gruppo SIEP-DIRECT'S. [Care across all phases of schizophrenia and initiation of treatment: discrepancy between routine practice and evidence. The SIEP-DIRECT'S Project]. Epidemiol Psichiatr Soc. 2008 Oct-Dec;17(4):305-18. Italian. PMID 19024719
- [Background] Ruggeri M, Lasalvia A, Bisoffi G, Thornicroft G, Vazquez-Barquero JL, Becker T, Knapp M, Knudsen HC, Schene A, Tansella M; EPSILON Study Group. Satisfaction with mental health services among people with schizophrenia in five European sites: results from the EPSILON Study. Schizophr Bull. 2003;29(2):229-45. doi: 10.1093/oxfordjournals.schbul.a007000. PMID 14552499
- [Background] Ruggeri M, Lasalvia A, Tansella M, Bonetto C, Abate M, Thornicroft G, Allevi L, Ognibene P. Heterogeneity of outcomes in schizophrenia. 3-year follow-up of treated prevalent cases. Br J Psychiatry. 2004 Jan;184:48-57. doi: 10.1192/bjp.184.1.48. PMID 14702227
- [Background] Semisa D, Casacchia M, Di Munzio W, Neri G, Buscaglia G, Burti L, Pucci C, Corlito G, Bacigalupi M, Parravani R, Roncone R, Cristofalo D, Lora A, Ruggeri M; Gruppo SIEP-DIRECT'S. [Promoting recovery of schizophrenic patients: discrepancy between routine practice and evidence. The SIEP-DIRECT'S Project]. Epidemiol Psichiatr Soc. 2008 Oct-Dec;17(4):331-48. Italian. PMID 19024721
- [Background] Community-based psychiatry: long-term patterns of care in South-Verona. Psychol Med Monogr Suppl. 1991;19:1-54. PMID 1745696
- [Background] Lasalvia A, Gentile B, Ruggeri M, Marcolin A, Nose F, Cappellari L, Lamonaca D, Toniolo E, Busana C, Campedelli A, Cuccato G, Danieli A, De Nardi F, De Nardo V, Destro E, Favaretto G, Frazzingaro S, Giacopuzzi M, Pristinger P, Pullia G, Rodighiero S, Tito P, Aprile F, Nicolaou S, Coppola G, Garzotto N, Gottardi U, Lazzarin E, Migliorini G, Pavan L, Ramaciotti F, Roveroni P, Russo S, Urbani P, Tansella M; Gruppo Picos-Veneto. [Heterogeneity of the Departments of Mental Health in the Veneto Region ten years after the National Plan 1994-96 for Mental Health. Which implication for clinical practice? Findings from the PICOS Project]. Epidemiol Psichiatr Soc. 2007 Jan-Mar;16(1):59-70. Italian. PMID 17427605
- [Background] Lasalvia A, Bonetto C, Bertani M, Bissoli S, Cristofalo D, Marrella G, Ceccato E, Cremonese C, De Rossi M, Lazzarotto L, Marangon V, Morandin I, Zucchetto M, Tansella M, Ruggeri M. Influence of perceived organisational factors on job burnout: survey of community mental health staff. Br J Psychiatry. 2009 Dec;195(6):537-44. doi: 10.1192/bjp.bp.108.060871. PMID 19949206
- [Derived] Espinosa R, Trucharte A, Contreras A, Peinado V, Valiente C. Who Benefits Most from Positive Psychological Interventions? Predictors and Moderators of Well-Being Outcomes in Severe Mental Health Conditions. Healthcare (Basel). 2025 Aug 13;13(16):1988. doi: 10.3390/healthcare13161988. PMID 40868604
- [Derived] Lasalvia A, Bonetto C, Lenzi J, Rucci P, Iozzino L, Cellini M, Comacchio C, Cristofalo D, D'Agostino A, de Girolamo G, De Santi K, Ghigi D, Leuci E, Miceli M, Meneghelli A, Pileggi F, Scarone S, Santonastaso P, Torresani S, Tosato S, Veronese A, Fioritti A, Ruggeri M; GET UP Group. Predictors and moderators of treatment outcome in patients receiving multi-element psychosocial intervention for early psychosis: results from the GET UP pragmatic cluster randomised controlled trial. Br J Psychiatry. 2017 May;210(5):342-349. doi: 10.1192/bjp.bp.116.190058. Epub 2017 Mar 16. PMID 28302703
- [Derived] Ruggeri M, Bonetto C, Lasalvia A, De Girolamo G, Fioritti A, Rucci P, Santonastaso P, Neri G, Pileggi F, Ghigi D, Miceli M, Scarone S, Cocchi A, Torresani S, Faravelli C, Zimmermann C, Meneghelli A, Cremonese C, Scocco P, Leuci E, Mazzi F, Gennarelli M, Brambilla P, Bissoli S, Bertani ME, Tosato S, De Santi K, Poli S, Cristofalo D, Tansella M; GET UP GROUP; Ruggeri M, Mirella ME, Bissoli S, Bonetto C, Cristofalo D, De Santi K, Lasalvia A, Lunardi S, Negretto V, Poli S, Tosato S, Zamboni MG, Ballarin M, De Girolamo G, Fioritti A, Neri G, Pileggi F, Rucci P, Bocchio Chiavetto L, Scasselatti C, Zanardini R, Brambilla P, Bellani M, Bertoldo A, Marinelli V, Negretto V, Perlini C, Rambaldelli G, Lasalvia A, Bertani M, Bissoli S, Lazzarotto L, Bardella S, Gardellin F, Lamonaca D, Lasalvia A, Lunardon M, Magnabosco R, Martucci M, Nicolau S, Nifosi F, Pavanati M, Rossi M, Piazza C, Piccione G, Sala A, Sale A, Stefan B, Zotos S, Balbo M, Boggian I, Ceccato E, Dall'Agnola R, Gardellin F, Girotto B, Goss C, Lamonaca D, Lasalvia A, Leoni R, Mai A, Pasqualini A, Pavanati M, Piazza C, Piccione G, Roccato S, Rossi A, Sale A, Strizzolo S, Zotos S, Urbani A, Ald F, Bianchi B, Cappellari P, Conti R, De Battisti L, Lazzarin E, Merlin S, Migliorini G, Pozzan T, Sarto L, Visona S, Brazzoli A, Campi A, Carmagnani R, Giambelli S, Gianella A, Lunardi L, Madaghiele D, Maestrelli P, Paiola L, Posteri E, Viola L, Zamberlan V, Zenari M, Tosato S, Zanoni M, Bonadonna G, Bonomo M, Santonastaso P, Cremonese C, Scocco P, Veronese A, Anderle P, Angelozz A, Amalric I, Baron G, Candeago EB, Castelli F, Chieco M, Cremonese C, Di Costanzo E, Derossi M, Doriguzzi M, Galvano O, Lattanz M, Lezzi R, Marcato M, Marcolin A, Marini F, Matranga M, Scalabrin D, Zucchetto M, Zadro F, Austoni G, Bianco M, Bordino F, Dario F, De Risio A, Gatto A, Grana S, Favero E, Franceschin A, Friederici S, Marangon V, Pascolo M, Ramon L, Scocco P, Veronese A, Zambolin S, Riolo R, Buffon A, Cremonese C, Di Bortolo E, Friederici S, Fortin S, Marcato M, Matarrese F, Mogni S, Codemo N, Russi A, Silvestro A, Turella E, Viel P, Dominoni A, Andreose L, Boemio M, Bressan L, Cabbia A, Canesso E, Cian R, Dal Piccol C, Dalla Pasqua MM, Di Prisco A, Mantellato L, Luison M, Morgante S, Santi M, Sacillotto M, Scabbio M, Sponga P, Sguotto ML, Stach F, Vettorato MG, Martinello G, Dassie F, Marino S, Cibiniel L, Masetto I, Marcato M, Cabianca O, Valente A, Caberlotto L, Passoni A, Flumian P, Daniel L, Gion M, Stanziale S, Alborino F, Bortolozzo V, Bacelle L, Bicciato L, Basso D, Navaglia F, Manoni F, Ercolin M, Neri G, Giubilini F, Imbesi M, Leuci E, Mazzi F, Semrov E, Giovanni CS, Taro e Ceno V, Ovest P, Anelli S, Amore M, Bigi L, Britta W, Anna GB, Bonatti U, Borziani M, Crosato I, Galluccio R, Galeotti M, Gozzi M, Greco V, Guagnini E, Pagani S, Maccherozzi M, Marchi F, Melato E, Mazzucchi E, Marzullo F, Pellegrini P, Petrolini N, Volta P, Anelli S, Bonara F, Brusamonti E, Croci R, Flamia I, Fontana F, Losi R, Mazzi F, Marchioro R, Pagani S, Raffaini L, Ruju L, Saginario A, Tondelli MG, Marrama D, Bernardelli L, Bonacini F, Florindo A, Merli M, Nappo P, Sola L, Tondelli O, Tonna M, Torre MT, Tosatti M, Venturelli G, Zampolla D, Bernardi A, Cavalli C, Cigala L, Ciraudo C, Di Bari A, Ferri L, Gombi F, Leurini S, Mandatelli E, Maccaferri S, Oroboncoide M, Pisa B, Ricci C, Poggi E, Zurlini C, Malpeli M, Colla R, Teodori E, Vecchia L, D'Andrea R, Trenti T, Paolini P, Mazzi F, Carpeggiani P, Pileggi F, Ghigi D, Gagliostro M, Pratelli M, Rucci P, Lazzaro S, Antonelli A, Battistini L, Bellini F, Bonini E, Capelli CB, DiDomizio C, Drei C, Fucci G, Gualandi A, Grazia MR, Losi AM, Mazzoni FM, Marangoni D, Monna G, Morselli M, Oggioni A, Oprandi S, Paganelli W, Passerini M, Piscitelli M, Reggiani G, Rossi G, Salvatori F, Trasforini S, Uslenghi C, Veggetti S, Bartolucci G, Baruffa R, Bellini F, Bertelli R, Borghi L, Ciavarella P, DiDomizio C, Monna G, Oggioni A, Paltrinieri E, Rizzardi F, Serra P, Suzzi D, Carlo U, Piscitelli M, Arienti P, Aureli F, Avanzi R, Callegari V, Corsino A, Host P, Michetti R, Pratelli M, Rizzo F, Simoncelli P, Soldati E, Succi E, Bertozzi M, Canetti E, Cavicchioli L, Ceccarelli E, Cenni S, Marzola G, Gallina V, Leoni C, Olivieri A, Piccolo E, Ravagli S, Russo R, Tedeschini D, Verenini M, Abram W, Granata V, Curcio A, Guerra G, Granini S, Natali L, Montanari E, Pasi F, Ventura U, Valenti S, Francesca M, Farneti R, Ravagli P, Floris R, Maroncelli O, Volpones G, Casali D, Miceli M, Bencini A, Cellini M, De Biase L, Barbara L, Charles L, Pratesi C, Tanini A, Cellini M, Miceli M, Loparrino R, Pratesi C, Ulivelli C, Cussoto C, Dei N, Fumanti E, Pantani M, Zeloni G, Bellini R, Cellesi R, Dorigo N, Gulli P, Ialeggio L, Pisanu M, Rinaldi G, Konze A, Cocchi A, Meneghelli A, Bianco M, Modignani L, Frova M, Monzani E, Zanobio A, Malagoli M, Pagani R, Barbera S, Morganti C, Monzani E, Amade ES, Brambilla V, Montanari A, Caterina G, Lopez C, Marocchi A, Moletta A, Sberna M, Cascio MT, Scarone S, Manzone ML, Barbara B, Mari L, Manzone ML, Razzini E, Bianchi Y, Pellizzer MR, Verdecchia A, Sferrazza MG, Manzone ML, Pismataro R, D'Eril GV, Barassi A, Pacciolla R, Faraci G, Torresani S, Rosmini B, Carpi F, Soelva M, Anderlan M, De Francesco M, Duregger E, Torresani S, Vettori C, Doimo S, Kompatscher E, Soelva M, Torresani S, Forer M, Kerschbaumer H, Gampe A, Nicoletti M, Acerbi C, Aquilino D, Azzali S, Bensi L, Bissoli S, Cappellari D, Casana E, Campagnola N, Dal Corso E, Di Micco E, Gobbi E, Ferri L, Gobbi E, Mairaghi L, Malak S, Mesiano L, Paterlini F, Perini M, Puliti EM, Rispoli R, Rizzo E, Sergenti C, Soave M, Alpi A, Bislenghi L, Bolis T, Colnaghi F, Fascendini S, Grignani S, Meneghelli A, Patelli G, Faravelli C, Casale S, Zimmermann C, Deledda G, Goss C, Mazzi M, Rimondini M, Gennarelli M, Scassellati C, Bonvicini C, Longo S, Bocchio Chiavetto L, Zanardini R, Ventriglia M, Squitti R, Frisoni G, Pievani M, Balestrieri M, Brambilla P, Perlini C, Marinelli V, Bellani M, Rambaldelli G, Bertoldo A, Atzori M, Mazzi F, Carpeggiani P, Beltramello A, Alessandrini F, Pizzini F, Zoccatelli G, Sberna M, Konze A, Politi P, Emanuele E, Brondino N, Martino G, Bergami A, Zarbo R, Riva MA, Fumagalli F, Molteni R, Calabrese F, Guidotti G, Luoni A, Macchi F, Artioli S, Baldetti M, Bizzocchi M, Bolzon D, Bonello E, Cacciari G, Carraresi C, Cascio MT, Caselli G, Furlato K, Garlassi S, Gavarini A, Lunardi S, Macchetti F, Marteddu V, Plebiscita G, Poli S, Totaro S, Bebbington P, Birchwood M, Dazzan P, Kuipers E, Thornicroft G, Pariante C, Lawrie S, Pariante C, Soares JC. A multi-element psychosocial intervention for early psychosis (GET UP PIANO TRIAL) conducted in a catchment area of 10 million inhabitants: study protocol for a pragmatic cluster randomized controlled trial. Trials. 2012 May 30;13:73. doi: 10.1186/1745-6215-13-73. PMID 22647399